CLINICAL TRIAL: NCT04634565
Title: A SINGLE CENTER, OPEN LABEL, SINGLE ARM STUDY TO INVESTIGATE THE REPEATED DOSE (FOR 10 DAYS) PHARMACOKINETICS AFTER ORAL ADMINISTRATION OF 200 MG PF-06651600 IN CHINESE HEALTHY ADULT PARTICIPANTS
Brief Title: PHARMACOKINETIC CHARACTERIZATION OF PF-06651600 IN CHINESE ADULT PARTICIPANTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B7981036
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-06651600 (Experimental): PF-06651600 200 milligrams(mg) once daily for 10 days
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — oral PF-06651600 tablet 200 mg once daily

SUMMARY:
This is an open label, single arm study in healthy Chinese male and/or female adult participants. Approximately 9 participants total are planned to participate in this study to ensure that a total of 8 evaluable participants (with all primary PK parameters) can complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Only females of non-childbearing potential
* Male and female Chinese participants who are healthy as determined by medical evaluation including a detailed medical history, complete physical examination, which includes blood pressure (BP) and pulse rate measurement, clinical laboratory tests, and 12 lead ECG.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 19 to 27 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg. Gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C, or syphilis; positive testing for HIV, hepatitis B, hepatitis C, and serological reaction of syphilis. Infection with hepatitis B or hepatitis C viruses according to protocol specific testing algorithm.
* Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline.
* History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
* Previous administration of an investigational drug within 90 days or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Single dose: maximum observed concentration (Cmax) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: time to reach maximum concentration (Tmax) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: area under the concentration-time curve from time 0 to infinity (AUCinf) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: area under the concentration-time curve from time 0 to the time of last quantifiable concentration (AUClast) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: terminal half life (t1/2) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose:AUC24 | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: mean residence time (MRT) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: apparent volume of distribution (Vz/F) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Single dose: apparent oral clearance (CL/F) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day1
Multiple Dose: Cmax | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: Tmax | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: AUCtau (tau = 24 hours) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: t1/2 | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: accumulation ratio on AUCtau (Rac) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: accumulation ratio on Cmax(Rac, Cmax) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: lowest concentration observed during the dosing interval (Cmin) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: average concentration at steady state (Cav) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: MRT | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: apparent volume of distribution at steady state (Vss/F) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: CL/F | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: peak trough fluctuation (PTF) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: peak trough swing (PTS) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Multiple Dose: predicted accumulation ratio to estimate linearity (Rss) | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 16 and 24 hours after dosing on Day10
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | From Day1 till Day17
Number of participants with clinically significant change in vital signs from Baseline | From Day1 till Day17
Number of participants with clinically significant abnormalities in 12-lead electrocardiograms (ECGs) | From Day1 till Day17
Number of participants with clinically significant abnormalities in physical examination findings | From Day1 till Day17

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - North District of Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981036